CLINICAL TRIAL: NCT03639675
Title: A Single-arm, Non-randomized and Open-label Phase 3 Study Evaluating the Efficacy, Safety and Tolerability of Intravitreal Aflibercept in Japanese Patients With Neovascular Glaucoma (NVG)
Brief Title: Study to Learn How the Drug Aflibercept Works in in Japanese Patients With Increased Eye Pressure That is Caused by New Blood Vessels Growing in the Eye (Neovascular Glaucoma or NVG). Safety of the Drug and Patients' Tolerability of the Drug Injection is Also Studied
Acronym: VENERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19652
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2020-02-18 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma, Neovascular
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NVG patients (Experimental): Japanese patients with neovascular glaucoma
  Interventions: Drug: Aflibercept (EYLEA, BAY86-5321); Drug: Topical IOP-lowering drugs

INTERVENTIONS:
Drug: Aflibercept (EYLEA, BAY86-5321) — 2 mg (0.05 mL), Intravitreal injection (IVT), single dose.
Drug: Topical IOP-lowering drugs — A combination of at least 3 topical IOP-lowering drugs will be administered during a run-in phase before treatment and should be kept unchanged until IOP evaluation at Week 1, after which they may be reduced according to the investigator's opinion

SUMMARY:
The researchers in this trial want to learn how the drug aflibercept works in in Japanese patients with increased eye pressure that is caused by new blood vessels growing in the eye (neovascular glaucoma or NVG). They also want to find out how patient tolerate the application of the drug that is injected in the vitreous humor of the eye and if this will cause any medical problems during the trial (vitreous humor, also called vitreous body is the clear gel that fills the space between the lens and the retina of the eyeball).

ELIGIBILITY:
Inclusion Criteria:

* Japanese men and women aged 20 years or older
* Patients diagnosed as having NVG (neovascular glaucoma) with neovascularization in the anterior segment (both iris and anterior chamber angle)
* Patients with IOP (intraocular pressure) higher than 25 mmHg in the study eye due to anterior segment (both iris and anterior chamber angle) neovascularization

Exclusion Criteria:

* Patients with angle-closure due to conditions other than NVG or complete angle-closure due to NVG
* Patients with a known or suspected ocular or peri-ocular infection
* Patients with severe intraocular inflammation in the study eye
* Women who are pregnant, suspected of being pregnant or lactating
* Patients with known allergy to aflibercept

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - University of Fukui Hospital, Yoshida, Fukui
  - Tsukazaki Hospital, Himeji, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki, Osaka
  - Shimane University Hospital, Izumo, Shimane

REFERENCES:
- [Derived] Inatani M, Higashide T, Matsushita K, Nagasato D, Takagi H, Ueki M, Takai Y, Miyazaki K, Iwamoto Y, Kobayashi M, Leal S. Efficacy and Safety of Intravitreal Aflibercept Injection in Japanese Patients with Neovascular Glaucoma: Outcomes from the VENERA Study. Adv Ther. 2021 Feb;38(2):1106-1115. doi: 10.1007/s12325-020-01580-y. Epub 2020 Dec 16. PMID 33330959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 7 study sites in Japan from 3-Oct-2018 (first subject's first visit) to 14-Mar-2019 (last subject's last visit).
Pre-assignment Details: Overall, 17 participants were screened. Of these, 16 participants were assigned and received the study treatment.
Groups:
- Aflibercept 2 mg Intravitreal (IVT) Injection Group: Japanese patients with neovascular glaucoma
Period: Overall Study
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group
Started | 16
Received Treatment | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) From Baseline to Week 1
Description: The primary efficacy analysis was on the changes in IOP from baseline to Week 1 (LOCF).
Time Frame: Baseline and week 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group
Number analyzed (Participants) | 16
mmHg | -8.3 (7.3)
Statistical Analysis 1: Comparison: Aflibercept 2 mg Intravitreal (IVT) Injection Group; Test type: Other; p = 0.0004, one-sample t-statistics; Mean change = -8.3, 95% CI 2-sided [-12.2 to -4.4]

2. Secondary Outcome: Percentage of Participants Who Had Improved Neovascularization of the Iris (NVI) Grade From Baseline to Week 1
Description: NVI Grade: 0=No iris neovascularization; 1=Fine surface neovascularization of the pupillary zone of the iris involving less than two quadrants; 2=Surface neovascularization of the pupillary zone of the iris involving more than two quadrants; 3=In addition to neovascularization of the pupillary zone, neovascularization of the ciliary zone of the iris and/or ectropion uveae involving one to three quadrants; 4=In addition to neovascularization of the pupillary zone, neovascularization of the ciliary zone of the iris and/or ectropion uveae involving more than three quadrants. The change in NVI grades categorized to "Improved" means improvement by at least one grade from baseline.
Time Frame: Baseline and week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group
Number analyzed (Participants) | 16
Participants | 13

ADVERSE EVENTS:
Time Frame: 30 days from administration in each patients
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Intravitreal (IVT) Injection Group (N=16)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Intravitreal (IVT) Injection Group (N=16)
Corneal erosion (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 4 (4)
Eye pruritus (Eye disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period described in the contract with the head of the medical institution based on J-GCP (Good clinical practice). The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03639675/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT03639675/SAP_001.pdf